CLINICAL TRIAL: NCT06307301
Title: A Phase I Trial to Evaluate Safety and Tolerability of Abatacept Followed by Subcutaneous Interleukin-2 Administration in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Study in ALS With Abatacept & IL-2
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00031998
Record Dates: First submitted 2023-12-26; First posted 2024-03-12 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Abatacept; aldesleukin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase I Study in ALS with Abatacept & IL-2 (Experimental): Primary Objective:
  1. To assess the safety and the tolerability of abatacept followed by IL-2 administration in ALS patients
  Secondary Objectives:
  1. To investigate the immunomodulatory effects of abatacept followed by IL-2, by monitoring the change in the number of Tregs
  2. To investigate the immunomodulatory effects of abatacept followed by IL-2, by monitoring the change in the suppressive activity of Tregs on T effector proliferation.
  3. To investigate the immunomodulatory effects of abatacept followed by IL-2, by monitoring in the level of cytokines secreted by PBMCs throughout the course of the study
  Exploratory Objective:
  1. To characterize the effects of abatacept followed by IL-2 on clinical outcome measures of ALS, including the Appel ALS Rating Scale (AALS) and ALS Functional Rating Scale-Revised (ALSFRS-R) scores, and the forced vital capacity (FVC) and maximum inspiratory pressure (MIP).
  Interventions: Drug: Abatacept Injection [Orencia] and Proleukin (aldesleukin)

INTERVENTIONS:
Drug: Abatacept Injection [Orencia] and Proleukin (aldesleukin) — Abatacept (Orencia®) and recombinant human IL-2 (aldesleukin). Patients will receive a fixed dose of subcutaneous abatacept (125 mg/mL) at day 1. Two weeks later (day 15), patients will receive the second dose of subcutaneous abatacept (125 mg/mL). In addition, patients will receive subcutaneous IL-2 (1x106units /day) for 5 days (days 15-19). If this treatment regimen is tolerated, patients will receive 28 further similar treatment courses of abatacept and IL-2 every two weeks.

SUMMARY:
In Amyotrophic Lateral Sclerosis (ALS), the reduction of regulatory T-lymphocyte (Treg) numbers and suppressive function correlates with rapid disease progression. The investigator completed a phase 1 study of infusions of expanded autologous Tregs in combination with subcutaneous IL-2 injections in ALS patients, which showed enhancement of Treg numbers and suppressive function in vivo. The enhanced Treg suppressive function correlated strongly with slowing and stabilization of disease progression. Drugs that enhance endogenous Treg numbers and suppressive function may also stabilize disease in ALS. This phase 1 study aims to determine whether the combination therapy of subcutaneous IL-2 and abatacept (Orencia®) is safe and well-tolerated in 6 patients with ALS, and whether the therapy enhances Treg numbers and suppressive function in vivo.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for initial enrollment on this study if they meet the following criteria at the time of screening:

1. Provided informed consent and authorized use of protected health information (PHI) in accordance with national and local patient privacy regulations.
2. ALS meeting El Escorial criteria for possible, probable, lab-supported probable, or definite ALS.
3. At least 18 years old.
4. Total bilirubin less than or equal to 1.5 mg/dL
5. Alanine aminotransferase level (ALT) less than or equal to five times normal, albumin greater than or equal to 3.0 gm/dL
6. Serum creatinine less than 1.5 mg/dL
7. Capable of complying with all study procedures, including the study drug delivery procedure, in the Investigator's opinion.
8. A family member or caretaker who is expected to be consistently available to administer both study drugs of abatacept and IL-2 if the participant is unable to do so.
9. On a stable regimen of riluzole for at least 30 days at the time of screening. If not on riluzole at the time of study entry, willing to refrain from initiation of the agent for the duration of the trial.
10. Patients on edaravone willing to refrain from taking edaravone on the same day as they will receive the abatacept injection for the duration of the trial. If not on edaravone at the time of study entry, willing to refrain from initiation of the agent for the duration of the trial.
11. Forced vital capacity (FVC) ≥50% of predicted capacity for age, height, and sex at screening, or receiving treatment with noninvasive ventilation if FVC < 50% of predicted for age, height, and sex at screening.

Exclusion Criteria:

Patients will be ineligible to participate if any of the following are true at the time of screening:

1. Serious, active bacterial, fungal, or viral infection, active or latent tuberculosis.
2. Tracheostomy.
3. Severe cardiac dysfunction defined as left ventricular ejection fraction <40% if an echocardiogram is medically indicated to clarify ongoing symptoms or EKG findings.; a history of non-controlled cardiac arrhythmias; history of cardiac tamponade; Unstable angina or MI in the last 3 months.
4. Hypersensitivity or allergy to IL-2 or abatacept.
5. History of bowel ischemia/perforation, or GI bleeding requiring surgery.
6. History of resistant seizures, history of coma or toxic psychosis lasting >48 hours.
7. Platelets <100,000/mm3; hematocrit <30%.
8. History of cancer in the past 5 years (except cutaneous Basal cell carcinoma or squamous cell carcinoma).
9. Hx of immunomodulation therapy including IL-2 or abatacept administration in the past 90 days.
10. Treatment with another investigational drug, biological agent, or device within 30 days or 5 half-lives of screening, whichever is longer.
11. If female, breastfeeding, known to be pregnant, planning to become pregnant during the study, or unwilling to use effective contraception for the duration of the trial and for 90 days after treatment.
12. If male of reproductive capacity, unwilling to use effective contraception for the duration of the trial and for 90 days after treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2024-10-17 (Estimated); Study Completion 2024-10-17 (Estimated)

PRIMARY OUTCOMES:
To evaluate adverse events and laboratory abnormalities to assess the safety and tolerability of abatacept followed by Interleukin 2 (IL-2) administration in ALS patients | 24 months
  Incidence and severity of AEs, including changes in laboratory values and vital signs.
  The investigator will determine whether safety and tolerability of abatacept followed by IL-2 administration are acceptable in order to proceed with the next phase. Safety and tolerability will be assessed throughout the study.

SECONDARY OUTCOMES:
Change in Regulatory T cells (Tregs) numbers in the blood from baseline | Baseline to Week 15
  The change in the number of Tregs.will be monitored
  The investigator hypothesizes that increasing Treg numbers and suppressive function will slow the progression of ALS, and the investigator will determine whether these markers increase in response to Abatacept/IL-2 administration.
Change in Regulatory T cells (Tregs) suppressive function in the blood from baseline | Baseline to Week 15
  The change in the suppressive activity of Tregs on responder T cell proliferation will be monitored
  The investigator hypothesizes that increasing Treg numbers and suppressive function will slow the progression of ALS, and the investigator will determine whether these markers increase in response to Abatacept/IL-2 administration.
Changes in the level of cytokines secreted by PBMCs from baseline | Baseline to Week 15
  The level of cytokines secreted by PBMCs throughout the course of the study
  The investigator hypothesizes that modulating peripheral inflammatory cytokines will slow the progression of ALS, and the investigator will determine whether these markers decrease in response to Abatacept/IL2 administration.

OTHER OUTCOMES:
Changes in Appel Amyotrophic Lateral Sclerosis rating scale ( AALS) slope | Baseline to Week 16
  Clinical outcome measures of ALS, including the Appel ALS Rating Scale (AALS)
  Appel ALS score, range 30 to 164; 30 is normal and 164 is maximum impairment
  Validated measures of ALS progression were chosen to begin collecting data on treatment efficacy.
Changes in Amyotrophic Lateral Sclerosis functional rating scale-revised (ALSFRS-R) slope | Baseline to Week 16
  Clinical outcome measures of ALS, including thed ALS Functional Rating Scale-Revised (ALSFRS-R) scores
  ALS Functional Rating Scale-Revised, range 0 to 48; 48 is normal and 0 is maximum impairment
  Validated measures of ALS progression were chosen to begin collecting data on treatment efficacy.
Changes in forced vital capacity (FVC) and maximum inspiratory pressure (MIP) scores | Baseline to Week 16
  Clinical outcome measures of ALS, including the forced vital capacity (FVC) measured in percent predicated capacity.
  Forced Vital Capacity, range 0 to 100 %; higher scores represent better function.
  Validated measures of ALS progression were chosen to begin collecting data on treatment efficacy.
Changes in maximum inspiratory pressure (MIP) scores | Baseline to Week 16
  Clinical outcome measures of ALS, including maximum inspiratory pressure (MIP)
  Maximal Inspiratory Pressure, range 0 to 120 cm H2O; higher scores represent better function
  Validated measures of ALS progression were chosen to begin collecting data on treatment efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Thonhoff, MD, PhD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Research Institute, Houston, Texas, United States

REFERENCES:
- [Derived] Thonhoff JR, Beers DR, Zhao W, Faridar A, Thome A, Wen S, Zhang A, Wang J, Appel SH. A phase 1 proof-of-concept study evaluating safety, tolerability, and biological marker responses with combination therapy of CTLA4-Ig and interleukin-2 in amyotrophic lateral sclerosis. Front Neurol. 2024 Jun 10;15:1415106. doi: 10.3389/fneur.2024.1415106. eCollection 2024. PMID 38915796